CLINICAL TRIAL: NCT06409364
Title: A Prospective, Blinded, Randomised Clinical Trial of Fludrocortisone Compared With Placebo in Critically Ill Patients Presenting With Aneurysmal Subarachnoid Haemorrhage
Brief Title: FLudrocortisone Administration in Aneurysmal Subarachnoid Haemorrhage
Acronym: FLASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The George Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TGI-CCP-35274; 2030936 (Other Grant/Funding Number: Australian government, Medical Research Future Fund (MRFF) 2023)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aSAH
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Fludrocortisone

STUDY DESIGN:
Intervention Model Description: A multi-centre, prospective, blinded, randomised clinical trial of fludrocortisone compared with placebo in patients presenting with aneurysmal subarachnoid haemorrhage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded participant, care provider, investigator and outcome assessors. Study drug and placebo identical in appearance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study drug (Experimental): Fludrocortisone Acetate 100ug Q6 hourly, given enterally for 14 days
  Interventions: Drug: Fludrocortisone
- Placebo (Placebo Comparator): Matched placebo tablet Q6 hourly, given enterally for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fludrocortisone — small white tablet containing 100mcg of fludrocortsone
  Other Names: Flurinef
  Arms: Study drug
Drug: Placebo — Matched placebo tablet,
  Arms: Placebo

SUMMARY:
A multi-centre, prospective, blinded, randomised clinical trial of fludrocortisone compared with placebo in patients presenting with aneurysmal subarachnoid haemorrhage.

The study aim is to determine if early administration of enteral fludrocortisone in aneurysmal subarachnoid haemorrhage reduce death and dependency at six months.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid haemorrhage (aSAH)is a devastating form of stroke, that predominately affects a younger age group. There are approximately 2000 cases per year in Australia, with the majority occurring in patients between 45 and 64 years of age and with a significant female preponderance. The burden of mortality of this condition is high; a review of 11,327 cases from 2000 to 2015 by our group revealed a mortality rate of 29% in patients who survived to hospital admission, with no annual improvement in that rate from 2003 onwards. Moreover, a substantial proportion of survivors from aSAH are left with residual neurological deficits. Persistent neurocognitive changes including deficits in memory, executive functioning and language, fatigue, depression and post-traumatic stress have been reported in survivors, resulting in lower than normal health related quality of life (HRQoL).

Cognitive impairment persists even in patients with supposedly good neurological recovery, with up to 40% of patients unable to return to their previous occupation. Data from our group support these findings, suggesting that approximately 50% of patients report at least a moderate disability six months after hospital discharge.

The healthcare costs associated with aSAH are substantial. In Australia and New Zealand, most patients with aSAH are admitted to an Intensive Care Unit (ICU), and have a median length of stay of 9 and 20 days in ICU and hospital, respectively. The median hospital cost for managing a patient with high grade aSAH is A$41,824 (interquartile range A$9,933-A$97,332); without considering the need for rehabilitation, ongoing care, and loss of earnings. Data from a single centre estimated total hospital costs over a ten year period for this cohort at $8.3 million; only 52 patients out of 139 survived hospitalisation. In contrast, a 14 day course of fludrocortisone costs just over A$12 compared with A$4800 for an occupied ICU bed day. A low cost intervention which reduced ICU stay and improved outcomes would therefore be anticipated to have a substantial economic benefit.

There are a number of complications associated with aSAH, of which hyponatraemia (defined as a serum sodium concentration <135mmol/L) is one of the most common with a reported prevalence of between 35% to 77%.7,8 The primary cause appears to be a salt wasting syndrome caused by secretion of natriuretic peptides and associated with large urine outputs and hypovolaemia. Hyponatraemia in the setting of aSAH is of particular concern, as it may exacerbate cerebral oedema and is also associated with an increased risk of cerebrovascular vasospasm and cerebral infarction, as well as a longer duration of ICU admission. Our group has recently completed a prospective analysis of 356 patients with aSAH from Australia and New Zealand and demonstrated that patients in whom the sodium concentration decreases over the ICU stay have a higher likelihood of a worse neurological outcome at 6-months compared to those patients in whom the sodium concentration remains steady.

Management of hyponatraemia in aSAH is complicated by the need to maintain a neutral fluid balance, as a reduced circulating blood volume is associated with an increased risk of cerebral vasospasm and delayed neurological deficit. Standard treatment comprises IV volume resuscitation and use of hypertonic saline solutions. These interventions require frequent blood tests, strict attention to fluid balance and central venous access, which can only be provided in ICU or high dependency units.

Fludrocortisone is a synthetic adrenocortical steroid possessing potent mineralocorticoid activity. In standard doses it produces significant sodium and fluid retention and increases urinary potassium excretion. It is currently only approved by the Therapeutic Goods Association for treatment of Addison's disease and salt losing adrenogenital syndrome and is priced at 20c per dose (100µg tablet).

There are two previous randomised trials which have examined the effect of fludrocortisone treatment on hyponatraemia and sodium balance in aSAH. Mori et al randomised 30 patients with aSAH and demonstrated that fludrocortisone significantly reduced urinary sodium excretion and reduced the incidence of hyponatraemia compared to standard management. Similar findings were noted in a study of 91 aSAH patients by Hasan et al, who also reported a lower incidence of cerebral ischaemia in the group that received fludrocortisone compared to standard treatment (22% vs 31% respectively, p=0.3). The trials were not blinded, and hyponatraemia was not an inclusion criterion. A more recent trial in the treatment of cerebral salt wasting secondary to tuberculous meningitis demonstrated that patients receiving fludrocortisone corrected their serum sodium concentration significantly faster than those who received placebo (4 days vs 15 days; p=0.004), and had a significantly lower incidence of deep border zone cerebral infarction (6% vs 33%, p=0.04).

Two systematic reviews have examined the role of fludrocortisone in preventing hyponatraemia and improving outcomes in aSAH. A Cochrane review published in 2005 identified the two previous trials of fludrocortisone in aSAH described above, both of which were performed over twenty years ago. A study using hydrocortisone (which also has mineralocorticoid action) was also included in the analysis. Mineralocorticoid treatment with fludrocortisone was reported to reduce the relative risk of delayed cerebral ischaemia (DCI); (RR 0.65; 95% CI 0.33-1.27) and of poor outcome; (RR 0.33;95% CI 0.03-3.20). A pooled estimate demonstrated that these treatments were associated with an increased rate of adverse effects; (RR 1.75;95% CI 1.03-2.95). However, this finding appeared to be generated mainly by the increased rate of hyperglycaemia in the hydrocortisone trial, whereas the two trials of fludrocortisone reported no increase in adverse effects. The authors concluded that participant numbers were too small to draw definitive conclusions on the efficacy of fludrocortisone and that further randomised controlled trials were required.

The second systematic review published in 2017 identified only one additional study of fludrocortisone to those in the 2005 analysis; this was however a before and after observational study, not a clinical trial. The authors identified that fludrocortisone treatment led to a reduction in hyponatremia, natriuresis and circulating volume contraction. There was no statistically significant effect of mineralocorticoid treatment on symptomatic vasospasm or DCI (RR 0.6; 95% CI 0.35-1.03), although the 95% CI were in favour of clinical benefit (Figure 2). The authors concluded the current evidence was not sufficient to determine the effect of fludrocortisone treatment because the included studies were underpowered, and that larger randomised trials were warranted.

The Neurocritical Care Society treatment guidelines for aSAH comment that fludrocortisone may be used for treatment of hyponatremia and/or hypovolaemia, but make no recommendation for its use in prevention. It appears to be safe and well tolerated - anticipated adverse effects include hypokalaemia, hypertension and pulmonary oedema, but these appear to be rare. Mori et al reported an increased incidence of transient hypokalaemia. Hasan et al noted 4 episodes of pulmonary oedema - 2 each in the fludrocortisone and control groups.

Although some clinical guidelines have suggested fludrocortisone as a potential treatment for hyponatremia in aSAH, it is not widely used; our observational data from Australasian ICUs has shown that less than 10% of the patient cohort were prescribed fludrocortisone. Of note, these patients had better functional outcomes at six months. The likely reason for the lack of widespread adoption into clinical practice is that the trials by Mori and Hasan discussed above were small, unblinded, and published over twenty years ago. Not only has management of aSAH substantially changed in that time period, but neither trial was sufficiently powered to detect improvements in patient centred outcomes. The authors of the most recent meta-analysis concluded that the existing data did not reflect current practice, the trials were small, and so large prospective RCTs were required to confirm these findings.

Recent reviews have highlighted that fludrocortisone may be a useful adjunct in the treatment and prevention of hyponatremia in aSAH, but that the current evidence is insufficient to make treatment recommendations. Fludrocortisone therefore has the potential to prevent the onset of hyponatraemia in aSAH and lead to improved outcomes; this will be the first adequately designed trial to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosed with subarachnoid haemorrhage from an aneurysm confirmed on computed tomography angiography (CTA) or digital subtraction angiography (DSA) of the intra-cranial arteries
3. Aneurysm has been secured
4. Hospital admission for aSAH within 96 hours
5. Currently being treated in a critical care environment

Exclusion Criteria:

1. Unable to receive enteral medications
2. Pre-existing glucocorticoid or mineralocorticoid treatment
3. Previous allergic reaction to fludrocortisone
4. History of cardiac, hepatic, or renal failure
5. Hypernatremia or hyponatremia (Na>145mmol/L or Na<125mmol/L) on the most recent blood sample at the time of screening.
6. Death deemed imminent or inevitable
7. Pregnancy (confirmed or suspected)
8. Previous inclusion in the FLASH trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | Six months after randomisation
  The primary outcome measure will be the modified Rankin Scale (mRS) score. Scores range from 0-5 with 0 is no disability and 5 is severe.

SECONDARY OUTCOMES:
Subarachnoid Haemorrhage Outcome Tool (SAHOT) | Six months after randomisation
  The secondary outcome measure will be the Subarachnoid Haemorrhage Outcome Tool (SAHOT) score. Fifty-six questions, possible score 0-2, maximum total score = 112.

OTHER OUTCOMES:
mortality | 90 days
  90-day mortality
Major disability or death (Modified Rankin Score (mRS) or >=3) | 90 days
  Major disability or death at day 90 (mRS>=3). Scores range from 0-5 with 0 is no disability and 5 is severe. to meet this outcome the mRS >=3.
Days alive and free of ICU | 90 days
  Days alive and free of ICU
  Days alive and free of ICU from randomisation to 90 days
Days alive and at home | 90 days
  Number of days alive and free of ICU
Incidence of readmission to ICU | 90 days
  Incidence of readmission to ICU
Incidence of radiologically confirmed cerebral infarction | 90 days
  Incidence of radiologically confirmed cerebral infarction
Incidence of aneurysm rebleeding | 90 days
  Incidence of aneurysm rebleeding
Incidence of hydrocephalus | 90 days
  Incidence of hydrocephalus
World Health Organisation Disability Assessment Schedule (WHODAS) at 90 days post randomisation | 90 days
  WHO Disability Assessment Schedule (WHODAS) at 90 days post randomisation. The scoring has three steps: Step 1 - Summing of recoded item scores within each domain. Step 2 - Summing of all six domain scores. Step 3 - Converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
Quality of life survey at 90 days post randomisation | 90 days
  EQ-5D-5L at 90 days post randomisation. descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Incidence of hypokalaemia | 90 days
  number of hypokalaemia episodes
Incidence of hypernatraemia | 90 days
  number of incidences of hypernatraemia
Incidence of fluid overload | 90 days
  number of incidences of fluid overload

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Cohen, MBBS, Principal Investigator — Royal Brisbane Hospital, Brisbane, Australia; Anthony Delaney, MBBS, Principal Investigator — Royal North Shore Hospital, Sydney, Australia; Torg Westerlund, MBBS, Principal Investigator — John Hunter Hospital, Newcastle, Australia; Andrew Udy, BHB MB ChB, Principal Investigator — The Alfred Hospital, Melbourne, Australia; Alex Nesbitt, MBBS, Principal Investigator — Princess Alexandra Hospital; Ian Sepppelt, MBBS, Principal Investigator — Nepean Blue Mountains Local Health District; Mak Wei-Yun, MBBS, Principal Investigator — Monash Medical Centre; David Bowen, MBBS, Principal Investigator — Westmead Hospital; James McCulloch, MBChB, Principal Investigator — Gold Coast University Hospital; Humphrey Walker, MBBS, Principal Investigator — St Vincent's Hospital Melbourne; Sananta Dash, MBBS, Principal Investigator — Townsville University Hospital; Matthew MacPartlin, MBBS, Principal Investigator — Wollongong Hospital; Andrew Turner, MBBS, Principal Investigator — Royal Hobart Hospital; Gavin Salt, MBBS, Principal Investigator — Prince of Wales Hospital; Laura Tincknell, MBBS, Principal Investigator — Auckland City Hospital; Jason Wright, MBBS, Principal Investigator — Wellington City Hospital
Locations (16):
- Australia (14):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Brisbane Women's Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital (Melbourne), Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: Yes
Proposed RNA analysis sub-study
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Cohen J, Delaney A, Udy A, Andersen C, Anderson CS, Bellapart J, Burrell LM, Devaux A, Evans DM, Fitzgerald E, Garside T, Hammond N, Hardie M, Jeffree RL, Knowles S, Lassig-Smith M, Li Q, Nethathe G, Rajbhandari D, Ramanan M, Talbot P, Taylor C, Wright J, Young MJ, Young PJ, Venkatesh B. Fludrocortisone to treat patients with aneurysmal subarachnoid haemorrhage: Protocol for an international, phase 3, randomised, placebo-controlled, multicentre trial. Crit Care Resusc. 2025 Jun 30;27(2):100116. doi: 10.1016/j.ccrj.2025.100116. eCollection 2025 Jun. PMID 40677678